CLINICAL TRIAL: NCT02835573
Title: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Brief Title: Potential Diagnostic and Prognostic Value of microRNAs for the Patients of Sepsis-induced Myocardial Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Bin He, M.D./Ph.D., Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-018
Record Dates: First submitted 2016-07-11; First posted 2016-07-18 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Sepsis-induced Myocardial Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis-induced myocardial injury group: Patients admitted to the hospital with the diagnosis of Sepsis-induced myocardial injury
- Blank control group: Patients admitted to the hospital without the diagnosis of Sepsis-induced myocardial injury

SUMMARY:
The purpose of this study is to evaluate the potential diagnostic and prognosis value of circulating microRNAs compared with cTnI for the patients of sepsis-induced myocardial injury at the emergency department (ED) and intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sepsis:SOFA score increase >=2 at baseline level induced by infection.
2. Suspected myocardial injury,including 1 as follows at least:Low blood pressure or using vasoactive drugs; ECG changes(ST segment changes or pathological Q wave); Troponin elevation(> 0.5 μg/L); BNP elevation(> 4670pg/ml); Echocardiography: cardiac function decline(EF<50%).

Exclusion Criteria:

1. Skeletal muscle damage (induced by orthopedics, vascular surgery or trauma surgical disease, surgery);
2. Pregnant and lactating women;
3. Patients with mental disorders;
4. Patients are using other experimental drugs;
5. Refusal to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of sepsis-induced myocardial injury
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of microRNAs evaluate by qPCR in patients of sepsis-induced myocardial injury | Day 7

SECONDARY OUTCOMES:
Prognostic value of microRNAs in patients of sepsis-induced myocardial injury | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided